CLINICAL TRIAL: NCT04734925
Title: Study of the Impact of an Intervention Performed by a Clinical Pharmacist on Patients at Risk of Pneumococcal Infection at the End of Hospitalization
Acronym: IP-VAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2019/DF-01
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Vaccination
Keywords: antipneumococcal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In France, Streptococcus pneumoniae is the leading agent involved in community-acquired bacterial pneumopathies and bacterial meningitis. The frequency of these infections is increasing in at-risk subjects. Paradoxically, pneumococcal vaccination coverage in this type of patient is limited at the national level, even though the French High Council for Public Health (HCSP) has been extending the 13-valent conjugate and 23-valent non-conjugate double vaccination in this target population since March 2017.

These patients generally benefit from regular medical follow-up involving several health professionals in hospital or outpatient clinics. In spite of this, one of the factors identified as a hindrance to pneumococcal vaccination is the absence of a proposal from the doctor.

We would like to assess compliance with the recommendations for pneumococcal vaccination according to the High Council of Public Health (HCSP) in at-risk patients leaving hospital. We also wish to measure the potential impact of an intervention by the clinical pharmacist on the application of these recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in one of the departments participating in the study
* At risk of pneumococcal infection according to HCSP recommendations (1)
* Negative pneumococcal vaccination status
* Adult patient (≥18 years old)

Exclusion Criteria:

* Under safeguard of justice
* Unable to receive informed information
* Patient having objected to the use of their data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in the Vascular Surgery and Pneumology Departments of Nimes University Hospital
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
vaccine protocols dispensed by dispensing pharmacists. | 3 month
  number of vaccine protocols

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nimes, Nîmes, France

REFERENCES:
- [Result] Chiappin M, Leguelinel-Blache G, Roux-Marson C, Kinowski JM, Dubois F. Impact of a clinical pharmacist's intervention on pneumococcal vaccination in a population of at- risk hospitalized patients: The IP-VAC study. Infect Dis Now. 2023 Oct;53(8):104765. doi: 10.1016/j.idnow.2023.104765. Epub 2023 Jul 25. PMID 37499757